CLINICAL TRIAL: NCT05237973
Title: Investigational Use of Neuromuscular Ultrasound
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000625; 000625-N
Record Dates: First submitted 2022-02-09; First posted 2022-02-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01-09

CONDITIONS: Muscular Dystrophy; Peripheral Neuropathy; Motor Neuron Disorder; Normal Physiology
Keywords: Neuromuscular; Ultrasound; Elastography; Muscle; Nerve; Natural History
MeSH Terms: conditions — Muscular Dystrophies; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuromuscular disorders: Diagnosed with a neuromuscular disorder such as motor neuron disorder, myopathy or have findings consistent with a peripheral neuropathy.
- Normal volunteers: No known abnormal muscle or nerve disorders

SUMMARY:
Background:

Current techniques used to measure the health and function of a person s nerves and muscles are generally effective, but they do have limits. Researchers are looking for ways to improve the ability to observe nerves and muscles and how they function in this natural history protocol.

Objective:

To study the use of ultrasound (sound waves) to learn more about nerves and muscles.

Eligibility:

Healthy adults, aged 18 and older, with no history of stroke, nerve or muscular disorders, or spine surgery are also needed. A smaller population of adults aged 18 and older who have a neuromuscular disorder or show symptoms of nerve or muscle disorder will also be evaluated.

Design:

Participants will be screened with a medical record review.

Participants will have up to 5 outpatient clinic visits. Most participants will have 1 or 2 visits. Visits will last for less than 3-4 hours each.

During each visit, participants will give a brief medical history and have a physical exam.

Participants will have ultrasounds to get pictures and measurements of their nerves and muscles. Gel will be applied to their skin. A probe will be placed on the skin surface. Sound waves sent through the probe will be used to create pictures.

Participants may have nerve conduction studies. Wires will be taped to the skin surface near a muscle or nerve in the arm or leg. The nerve will be stimulated with a small electric current that feels like a rubber band flick. The response will be recorded through the wires.

DETAILED DESCRIPTION:
Study Description:

Currently there are a limited number of biomarkers that can provide quantitative, reliable information about nerve and muscle function and structure in patients with neuromuscular diseases. This protocol aims to investigate and define specific ultrasound imaging techniques of nerves and muscles that may be useful as biomarkers in clinical trials. For nerve studies, we aim to evaluate the use of high resolution ultrasound probes for B-mode imaging including cross sectional area, diameter and nerve fascicle counts. Additional imaging modalities will be evaluated including shear wave elastography and low flow microvascular imaging. Ultrasound modalities for muscle imaging will include B-mode imaging, muscle thickness, echo-intensity and or shear wave imaging and low flow microvascular imaging. The hypothesis for incorporating these ultrasound imaging modalities into neuromuscular evaluations is these techniques can provide unique quantitative, reproducible data about the structure of nerves and muscles. This information can be used to compare patients with controls and measure change in these modalities in neuromuscular disease states and determine if these measures can serve as a reliable biomarker in neuromuscular diseases.

Objectives:

Primary Objectives:

* To acquire normative values for elastography of muscle in a population of healthy volunteers
* To acquire normative values for elastography of nerve in a population of healthy volunteers
* To acquire normative values of nerve fascicular count in a population of healthy volunteers
* To collect normal values of M-mode diaphragm imaging during quiet and deep breathing and voluntary sniff testing in a population of health controls to establish normal values.

Secondary Objectives:

* To determine the reproducibility of specialized techniques involving ultrasound of muscle and nerve: shear wave elastography in muscles and nerves, nerve fascicle counts
* To determine the presence or absence of low flow microvascular flow within nerves of a population of healthy volunteers

Exploratory Objectives:

* To compare shear wave elastography values (kPa, meters/second) with standard nerve conduction values; amplitude and nerve conduction velocities in healthy controls and participants with neuromuscular diseases.
* To compare shear wave elastography values with muscle thickness, echotexture and Heckmatt Scale values
* To compare shear wave elastography values (kPa, meters/second), nerve fascicle count and microvascular flow between volunteers with participants with neuromuscular disorders
* To compare B-mode quantitative measures of muscle in healthy controls and participants with neuromuscular diseases.
* To compare M-mode imaging values of diaphragm (excursion of movement) during quiet and deep breathing and voluntary sniff tests in healthy controls and patients with neuromuscular diseases.
* To quantitate the low flow microvascularity in nerves and muscles in healthy volunteers
* To develop a method for automated analysis of peripheral nerves that would allow for reproducible and refined imaging of nerves.

Endpoints:

Primary Endpoint:

* Muscle (deltoid, triceps, bicep, flexor carpi radialis, extensor digitorum communis, first dorsal interossei, rectus femoris, semimembranosus, tibialis anterior, medial gastrocnemius)elastography (m/s)
* Nerve (median and ulnar in the forearm, tibial in the calf) elastography (m/s)
* Nerve fascicular count (median and ulnar at wrist, tibial at ankle) in a population of normal volunteers (binary)
* M-mode diaphragm imaging during quiet and deep breathing and voluntary sniff testing in a population of health volunteers

Secondary Endpoints:

* Reproducibility

  * Muscle elastography (m/s)
  * Nerve elastography (m/s)
  * Nerve fascicle counts (#)
* Presence of low flow microvascularity in nerves (binary value)

Exploratory Endpoint:

* Amplitude (mV) and conduction velocity (m/s) obtained from standard nerve conduction studies and nerve elastography values (m/s) obtained from specialized techniques (median, ulnar, tibial)
* Ultrasound data on muscle thickness (mm) and Heckmatt Scale values (1-4)
* Nerve elastography (m/s), fascicular count (#), and microvascular flow (binary-yes/no)
* Muscle elastography (m/s), thickness (mm), Heckmatt scale
* M-mode imaging values of diaphragm (excursion of movement) during quiet and deep breathing and voluntary sniff tests
* Quantitative values of low flow microvascularity in muscles and nerves
* Reproducible ability to identify nerve and/or nerve associated structures using automated analysis

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Healthy Volunteers-Adults

   1. Healthy adults, male or female, aged 18 years old or older,
   2. In good general health as evidenced by medical history, medical conditions under control such as hypertension acceptable.
   3. Stated willingness to comply with all study procedures and availability for the duration of the study.
   4. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Participants with neuromuscular disorders

   1. Adults, male or female, aged 18 years old or older,
   2. Diagnosed with a neuromuscular disorder or have signs and symptoms of nerve or muscle disorder or neuromuscular diaphragm dysfunction.
   3. Stated willingness to comply with all study procedures and availability for the duration of the study.
   4. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Healthy Volunteers-Adults

   History of stroke, muscle disorders, peripheral neuropathy, or spine surgery
2. Participants with neuromuscular disorders

No clinical evidence of a neuromuscular disorder on clinical evaluation.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community and participants on other NIH protocols that have neuromuscular disorders.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
To collect normal values of M-mode diaphragm imaging during quiet and deep breathing and voluntary sniff testing in a population of health controls to establish normal values. | ongoing
  Normative values for M-mode imaging of the diaphragm in a population of healthy controls.
To acquire normative values for B-mode imaging of nerves (fascicle count) and muscles (quantitative echotexture measurement) and shear wave elastography data on muscle and nerve stiffness/speed of sound in a population of healthy volunteers. | ongoing
  Normative values for muscle and nerve shear wave elastography in a population of normal volunteers Normative values for nerve fascicular count in a population of normal volunteers

SECONDARY OUTCOMES:
To determine the reproducibility of specialized techniques involving ultrasound of muscle and nerve: shear wave elastography in muscles and nerves, nerve fascicle counts | ongoing
  Reproducibility of muscle and nerve shear wave elastography (meters/sec or kPa ) Reproducibility of nerve fascicle counts
To determine the presence or absence of low flow microvascular flow within nerves of a population of healthy volunteers | ongoing
  Presence of low flow microvascularity in nerves in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Tanya J Lehky, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Specific plan to make the IPD has not be made. This will have to be considered if the data is involved in a publication or other larger analysis.

REFERENCES:
- [Background] Creze M, Nordez A, Soubeyrand M, Rocher L, Maitre X, Bellin MF. Shear wave sonoelastography of skeletal muscle: basic principles, biomechanical concepts, clinical applications, and future perspectives. Skeletal Radiol. 2018 Apr;47(4):457-471. doi: 10.1007/s00256-017-2843-y. Epub 2017 Dec 9. PMID 29224123
- [Background] Saade DN, Neuhaus SB, Foley AR, Bonnemann CG. The Use of Muscle Ultrasound in the Diagnosis and Differential Diagnosis of Congenital Disorders of Muscle in the Age of Next Generation Genetics. Semin Pediatr Neurol. 2019 Apr;29:44-54. doi: 10.1016/j.spen.2019.01.001. Epub 2019 Jan 16. PMID 31060725
- [Background] Hobson-Webb LD. Emerging technologies in neuromuscular ultrasound. Muscle Nerve. 2020 Jun;61(6):719-725. doi: 10.1002/mus.26819. PMID 32012298
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000625-N.html